CLINICAL TRIAL: NCT05618678
Title: Pilot Testing Decision Making in Aging and Dementia for Autonomy for Preference-Based Care in Nursing Homes
Brief Title: Pilot Testing Decision Making in Aging and Dementia for Autonomy Program in Nursing Homes
Acronym: DIGNITY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Liza Behrens, PhD, RN, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00020594
Record Dates: First submitted 2022-09-22; First posted 2022-11-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Dementia; Staff Attitude; Nurse's Role; Nursing Homes
Keywords: Shared Decision Making; Person-Centered Care
MeSH Terms: conditions — Dementia | interventions — Infection Control

STUDY DESIGN:
Intervention Model Description: Nursing homes are randomized to one of two groups: 1.) DIGNITY Intervention (Protocol Manual, Baseline Education, ECHO Coaching) or 2.) Control Arm - (Infection Control Training - CDC Guidelines, Baseline Education, ECHO Coaching)
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not be aware of the randomization arm of the NH they are collecting data in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infection Control Training (Active Comparator): Nursing homes randomized to this arm of the study receive CDC guidelines and evidence based information on infection prevention prevention and control. Nursing home staff implement these standard in everyday resident care. Additionally, nursing home staff are invited to participate in Extension for Community Healthcare Outcomes (ECHO) sessions via real-time interactive videoconferencing software to support the implementation of the CDC guidelines and evidence-based practices.
  Interventions: Behavioral: Infection Control
- DIGNITY Intervention (Experimental): Nursing homes randomized to this arm of the study receive an evidence based risk assessment and care planning protocol for supporting decision making and aging in dementia for autonomy (DIGNITY). Nursing home staff use this manual to implement risk assessment and care planning for resident preferences that they perceive to carry a risk to the resident's health and/or safety. In addition nursing home staff participate in Extension for Community Healthcare Outcomes (ECHO) sessions via real-time interactive videoconferencing software to support the implementation of the DIGNITY protocol.
  Interventions: Behavioral: DIGNITY

INTERVENTIONS:
Behavioral: DIGNITY — DIGNITY is a multi-component, multi-level intervention that guides shared decision-making in nursing homes to support person-centered dementia care. Based in theory, this intervention targets nursing home staff attitudes and behaviors around assessing and judging whether to engage in risk situations to support resident preferences for everyday living and care despite cognitive decline due to dementia. It includes a protocol manual, baseline training on how to implement the DIGNITY strategy, and six ECHO sessions to help frontline staff negotiate intrinsic and cultural factors in preference situations that carry a risk to residents' health and safety.
  Arms: DIGNITY Intervention
Behavioral: Infection Control — This is an attention control intervention with similar dose of educational content and attention from interventionist. It includes distribution of links to the CDC Infection Control Practice Guidelines for nursing homes, a baseline training on infection control practices for frontline workers, and six ECHO coaching sessions.
  Arms: Infection Control Training

SUMMARY:
The purpose of this study is to adapt, pilot test, and evaluate the feasibility, acceptability, and preliminary effectiveness of DIGNITY (Decision-making In aGing and demeNtIa for auTonomY) for Preference-Based Care in Nursing Homes as a new evidence-based intervention to support nursing home staff to safely honor care and activity preferences of residents' living with dementia in rural, typically under resourced nursing home communities.

DETAILED DESCRIPTION:
Of 6.5 million older Americans are living with Alzheimer's disease and related forms of dementia (ADRD), two thirds will die in a nursing home (NH) where staff are not prepared to deliver a minimal level of federally mandated care. Care in NHs is delivered by an ever-changing workforce of 1.3 million staff members who are responsible to provide person-centered care (PCC)- that is care based on knowing and honoring residents preferences for care and activities of daily living. NH residents have reported they are not satisfied with efforts to honor their preferences for everyday living and care activities. For residents living with ADRD this can lead to a loss of dignity, anger, agitation, isolation, depression, and negative social interactions between residents ultimately reducing quality of life. A prominent, known barrier to honoring residents' preferences is the predominantly risk adverse attitudes and behaviors of NH staff. DIGNITY (Decision-making in aging and dementia for autonomy) is novel multi-level intervention based in theory and evidence aimed at empowering nursing home staff to negotiate residents' risky preferences by addressing intrinsic and system barriers to safely honoring a resident's preferences with decision aids, care planning, and staff coaching/education. In the proposed project, we will implement DIGNITY in a pilot cluster randomized trial of 120 nursing home staff and residents across four rural nursing homes located in Pennsylvania. Our aims are to: 1.) To explore stakeholder perspectives on the relevance and feasibility of implementing the DIGNITY intervention in rural, underserved nursing home communities; and 2.) examine the feasibility, acceptability, and preliminary effectiveness of DIGNITY within four rural, underserved nursing homes. Outcomes will be evaluated at baseline and 12 weeks following baseline education on the DIGNITY protocol. This study is a critical next step in developing evidence-based interventions that target gaps in direct-care workforce skills needed to enhance quality of care delivery to persons with ADRD living in NHs.

ELIGIBILITY:
Inclusion Criteria for Nursing Homes:

1. Located in rural Pennsylvania as defined by the Center for Rural Pennsylvania
2. Administrator articulates commitment to delivering person-centered care
3. NH has a dedicated dementia care unit and/or a total bed capacity of 50 beds or more
4. NH has the capacity to participate in the study activities for the term of the study as determined by nursing home leadership
5. NH has a dedicated quality improvement/safety team that meets regularly
6. NH has a stable internet connectivity for program delivery

Exclusion Criteria:

* Nursing Home does not meet inclusion criteria.

Convenience sampling will be used to recruit nursing home staff and residents within nursing homes.

Inclusion criteria for Nursing Home Staff:

1. 18 years or older
2. Employed by the participating nursing home for at least 6 months
3. Fluent in written and spoken English
4. Provides and/or influences direct care delivery to older adults with dementia

Inclusion criteria for Residents:

1. Resides in nursing home study site for at least 3 months
2. English speaking
3. Documented diagnosis of Alzheimer's disease or related dementia (ADRD)
4. Have a stated preference that nursing home staff indicated poses a risk to their health and/or safety
5. Provides consent/assent to be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Intervention Feasibility | 12 weeks after baseline education on DIGNITY protocol
  Evidence of Feasibility (Feasibility of Intervention Measure)
Staff Behavioral Intent | 12 weeks after baseline education on DIGNITY protocol
  Evidence of Staff Intent to Honor Resident's Preference (Investigator developed survey item)
Resident Satisfaction | 12 weeks after baseline education on DIGNITY protocol
  Evidence of resident satisfaction with preference (Preferences for Everyday Living Inventory)
Intervention Fidelity | 12 weeks after baseline education on DIGNITY protocol
  Evidence of staff fidelity to the DIGNTY Intervention (Investigator developed DIGNITY Intervention Fidelity Assessment Checklist)

SECONDARY OUTCOMES:
Staff Self - Efficacy | 12 weeks after baseline education on DIGNITY protocol
  Changes in perceived self-efficacy in Person-Centered Risk Management (Investigator Developed Self Efficacy Survey for Person-Centered Risk Management)
Intervention Acceptability | 12 Weeks after baseline education on DIGNITY protocol
  Staff rate intervention acceptability on the Acceptability of Intervention Measure

CONTACTS AND LOCATIONS:
Overall Officials: Liza Behrens, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No